CLINICAL TRIAL: NCT02537665
Title: Heating Precondition of Epidural Catheter Decrease the Incidence of Injury to Blood Vessel During Epidural Catheter Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Geng guiqi, PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19990807
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Epidural Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- incidence of bleeding (Other): the effect of the epidural catheter filled with heated or normal saline before inserting into epidural on the incidence of bleeding.
  Interventions: Other: heating precondition
- inserting time of catheter (Placebo Comparator): record the time from beginning of catheter inserting to completing the placement of the catheter.
  Interventions: Other: heating precondition

INTERVENTIONS:
Other: heating precondition

SUMMARY:
To explore the effect of heating precondition of epidural catheter on the incidence of injury to blood vessel during epidural catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery
* Epidural anesthesia.

Exclusion Criteria:

* blood coagulation disorders

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
the incidence of injury to blood vessel during epidural catheter placement | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China